CLINICAL TRIAL: NCT00260091
Title: Conventional Infertility Therapy vs. Fast Track to IVF
Brief Title: Conventional Infertility Treatment vs. Fast Track to IVF
Acronym: FASTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01HD038561 (NIH)
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2009-01

CONDITIONS: Infertility
Keywords: Infertility; Advanced maternal age; Pregnancy; Reproductive health; Fertility treatment; Reproduction
MeSH Terms: conditions — Infertility | interventions — Reproductive Techniques, Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I. (Active Comparator): Conventional infertility therapy
  Interventions: Procedure: intrauterine insemination; Procedure: infertility
- II. (Active Comparator): Fast track to in vitro fertilization therapy
  Interventions: Procedure: intrauterine insemination; Procedure: infertility

INTERVENTIONS:
Procedure: intrauterine insemination — An assisted reproduction technique which deposits washed sperm directly into the uterus, bypassing the cervix, and allowing the sperm to enter the fallopian tubes where fertilization normally occurs.
  Other Names: assisted reproductive technologies; IUI
Procedure: infertility — This procedure involves stimulating the ovaries, retrieving released eggs, fertilizing the eggs, growing the embryos in a laboratory, and then implanting the embryos in the woman's uterus to develop naturally.
  Other Names: assisted reproductive technologies

SUMMARY:
The purpose of this randomized prospective clinical trial is to determine whether an infertility treatment that moves quickly to In Vitro Fertilization (IVF) is more cost effective than the usual treatment strategy which includes various combinations of infertility drugs and intrauterine insemination (IUI) prior to utilizing In Vitro Fertilization.

DETAILED DESCRIPTION:
This is a randomized clinical trial to evaluate the efficacy, adverse events, and particularly cost and cost-effectiveness of two alternative infertility treatment strategies for patients who would otherwise be candidates for ovulation induction and IUI as their initial treatment. The two therapies compared are conventional treatment and fast track to IVF. Conventional therapy is a cost-conscious progressive treatment strategy that begins with the least invasive form of ovulation induction, clomiphene/IUI. It then progresses to FSH/IUI and, if pregnancy is not achieved, to IVF. The fast track to IVF strategy begins with clomiphene/IUI; if pregnancy does not result, these patients bypass FSH/IUI and move directly to IVF. We hypothesize that the fast track to IVF therapy results in a higher pregnancy rate, lower rates of medical complications during treatment, lower rates of pregnancy complications, and costs no more than conventional infertility treatment.

The trial has the following specific aims:

Aim 1: To compare the number of deliveries per initiated cycle, the proportion of women with a clinically recognized intrauterine pregnancy, and the time to clinical pregnancy between fast track to IVF and the conventional treatment arms of the clinical trial.

Aim 2: To compare the frequency of infertility treatment complications between the fast track to IVF arm and the conventional treatment arm.

Aim 3: To compare the occurrence of pregnancy complications between the fast track to IVF arm and the conventional treatment arm.

Aim 4: To evaluate the costs and cost effectiveness of the two alternative treatment strategies by comparing the direct and indirect medical costs between the fast track to IVF and conventional treatment arms of the clinical trial.

This is a collaborative study between Boston IVF, Harvard Vanguard Medical Associates, Harvard School of Public Health, Blue Cross Blue Shield of Massachusetts, Harvard Pilgrim Health Care, and Tufts Health Plan.

Total Enrollment: 503 Couples

ELIGIBILITY:
Inclusion Criteria:

* Female partner age 21 up to 40th birthday, at the time of recruitment. Infertility is defined as failure to conceive a recognized pregnancy after one year (or 12 menstrual cycles) of unprotected intercourse.
* Male partner has a normal semen analysis with a sperm concentration of >15 million total motile sperm, >1% normal forms by strict criteria, or >5 million total motile sperm on IUI prep.
* Female patient has at least one ovary and at least one ipsilateral patent fallopian tube confirmed by HSG or laparoscopy; pelvic pathology amenable to operative laparoscopy (pelvis restored to functional). The open tube cannot have had a previous ectopic (tubal) pregnancy and the closed tube cannot be a hydrosalpinx (a tube that is blocked at the end and filled with fluid), unless a tubal ligation has been performed at the junction of the uterus and fallopian tube.
* Patients with surgically corrected stages I and II endometriosis will be included.
* Normal uterine cavity demonstrated by HSG, Sonohysterogram (SHG), or hysteroscopy; pathologies of uterine cavity amenable to operative hysteroscopy (cavity restored to normal and demonstrated by post operative study).
* Anovulatory patients who did not conceive after a minimum of three ovulatory cycles with any medications, not including gonadotropin therapy. Anovulatory patients unable to achieve ovulation at dosages up to 150 mg of clomiphene or standard dosages of other ovulation inducing medications (i.e. bromocriptine). Hypoestrogenic hypothalamic amenorrhea patients will qualify immediately for inclusion, prior to any gonadotropin therapy.
* Normal ovarian reserve demonstrated in all patients i.e., cycle day 3 FSH/E2 values of <15 mIU/mL and <100 pg/mL, respectively. Normal TSH and prolactin.
* Female body mass index ≤ 38.

Exclusion Criteria:

* Previous tubal reconstructive surgery in which the pelvis was not restored to functional.
* Unilateral or bilateral hydrosalpinx (a tube that is blocked at the end and filled with fluid) that has not had a tubal ligation performed at the junction of the uterus and fallopian tubes.
* A laparoscopy that demonstrated pelvic adhesions or endometriosis for which the pelvis could not be restored to normal by surgery or endometriosis was not ablated or excised. All patients with stages III and IV endometriosis.
* One or more prior ectopic pregnancies in which one or both tubes were rendered nonfunctional; two or more ectopic pregnancies, even if tubes are patent.
* Severe male factor (i.e.; semen analysis with a sperm concentration of <15 million total motile sperm, <1% normal forms by strict criteria, or <5 million total motile sperm on IUI prep). Couples using donor semen will be excluded.
* Previous treatment with IUI or IVF. Previous treatment of normal ovulation patients with gonadotropins.
* Inadequate ovarian reserve demonstrating FSH >15 mIU/mL or estradiol > 100 pg/mL.
* Patients requiring gamete intrafallopian tube transfer (GIFT), zygote intrafallopian tube transfer (ZIFT), or tubal embryo transfer (TET).
* Female body mass index > 38.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 503 (Actual)
Dates: Start 1999-08; Primary Completion 2005-08 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Determine the cost-effectiveness of fast track to IVF versus conventional infertility treatment by conducting a randomized clinical trial to compare success rates and costs, as well as the associated complications of treatment. | at end of study

SECONDARY OUTCOMES:
Demographics and baseline variables will be collected, including: medical and reproductive history, age, education, income, race, nutritional history, smoking history, and clinical variables related to infertility diagnosis and treatment. | at end of study

CONTACTS AND LOCATIONS:
Overall Officials: Richard H. Reindollar, M.D., Principal Investigator — Dartmouth-Hitchcock Medical Center, Dartmouth Medical School, Lebanon, New Hampshire; Marlene B. Goldman, Sc.D., Study Director — Dartmouth-Hitchcock Medical Center
Locations (7):
- United States (7):
  - Harvard Vanguard Medical Associates, Boston, Massachusetts
  - Boston IVf, Brookline, Massachusetts
  - Harvard Vanguard Medical Associates, Burlington, Massachusetts
  - Boston IVF, Quincy, Massachusetts
  - Harvard Vanguard Medical Associates, Quincy, Massachusetts
  - Boston IVF, Waltham, Massachusetts
  - Harvard Vanguard Medical Associates, Wellesley, Massachusetts

REFERENCES:
- [Result] Goldman MB, Hartman TJ, Regan MM, Thornton KL, Neumann PJ, Alper MM, Reindollar RH. Dietary antioxidant status in couples with unexplained infertility: the fast track and standard treatment trial (FASTT). [abstract 361]. SGI, Los Angeles, California. J Soc Gynecol Inves 2005;12(2) Suppl:201A.
- [Result] Reindollar RH, Regan MM, Neumann PJ, Thornton KL, Alper MM, Goldman MB. A randomized controlled trial of 503 couples assigned to conventional infertility treatment or an accelerated track to IVF: Preliminary results of the Fast Track and Standard Treatment (FASTT) Trial [abstract O-108]. ASRM, Washington D.C. Fertil Steril 2007;88(1) Suppl:S41. (General Program Prize Paper Award)
- [Derived] Ruder EH, Hartman TJ, Reindollar RH, Goldman MB. Female dietary antioxidant intake and time to pregnancy among couples treated for unexplained infertility. Fertil Steril. 2014 Mar;101(3):759-66. doi: 10.1016/j.fertnstert.2013.11.008. Epub 2013 Dec 17. PMID 24355050